CLINICAL TRIAL: NCT03059069
Title: The Effect of Gliatamin (Chonline Alphoscerate) on Depressive Mood in Type 2 Diabetes Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2016-0349
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Type2 Diabetes With Depressive Mood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glitamin (Experimental): 800mg/day
  Interventions: Drug: Chonline Alphoscerate
- Placebo (Placebo Comparator): same shape, color, size tablet as Glitamin
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Chonline Alphoscerate — Patients treated with Chonline Alphoscerate as add on therapy to their medication
  Other Names: Gliatamin
  Arms: Glitamin
Drug: Placebo Oral Tablet — Patients maintain their medication with either Gliatamin or placebo for 6 months.
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of Gliatamin (chonline alphoscerate) on depressive mood in type 2 diabetes patients and demonstrate the impact of improved depressive mood could be influence the patient's quality of life and glycemic control.

DETAILED DESCRIPTION:
The prevalence of depressive disorder is higher in individuals with chronic diseases, and the screening and management of depression is emphasized. Diabetes mellitus (DM) is a class of chronic disease and the incidence of DM has been increasing. According to previous study, 31.1% of patients with DM accompanied with depressive disorders which was higher than that of subjects without DM. Furthermore, DM as well as depression is known for risk factor for dementia.

The choline metabolism involves in neuropathology of depressive disorders and individuals with depressive disorders showed the lower level of choline concentration. Choline alphoscerate is cholinergic precursor and showed the favorable clinical results in dementia management.

As pseudodementia can be presented as depressive disorder and choline alphoscerate would be an option for these cases. Therefore, the aim of this study is to investigate the effect of Gliatamin (chonline alphoscerate) on depressive mood in type 2 diabetes patients and demonstrate the impact of improved depressive mood could be influence the patient's quality of life and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Age ≥ 50
* Glycemic control: HbA1c ≤ 10.0%
* 10 ≤ Beck Depression Inventory (BDI) <30 points
* Participants who can undergo contraception in case of being in childbearing period
* Understands the study procedure, alternatives, and risks and voluntarily agrees to participate by giving written informed concent

Exclusion Criteria:

* Type 1 diabetes, Secondary diabetes, gestational diabetes
* Ongoing dementia treatment or anti-depressive disorder medication
* Uncontrolled psychiatric disorder
* BDI ≥ 30 points
* Heavy alcoholics
* Underlying chronic liver disease (hemochromatosis, liver cell carcinoma, autoimmune liver disease, liver cirrhosis, chronic viral hepatitis)
* Allergy or hypersensitivity to target medication or any of its components
* Renal failure, moderate or severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m2), or ongoing dialysis
* Abnormal liver function (AST/ALT > x3 upper normal limit)
* History of alcohol or drug abuse in the previous 3 months
* Premenopausal women who are nursing or pregnant
* Human immunodeficiency virus (HIV) or human immunodeficiency virus (AIDS)
* chronic pancreatitis or pancreatic cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
changes in Hamilton Depression Rating Scale (HDRS) | 6 months after the treatment
  The HDRS will be scored by face-to-face interview.

SECONDARY OUTCOMES:
changes in Mini-mental state examination (MMSE) score | 6 months after the treatment
  MMSE questionnaire will be checked by careful interview and self-reported.
glucometabolic parameters | 6 months after the treatment
  fasting glucose (mg/dL)
glucometabolic parameters | 6 months after the treatment
  postprandial 2h glucose (mg/dL)
glucometabolic parameters | 6 months after the treatment
  fasting insulin (uIU/mL)
glucometabolic parameters | 6 months after the treatment
  homeostasis model assessment for insulin resistance (mg/dL•uIU/mL)
glucometabolic parameters | 6 months after the treatment
  aspartate aminotransferase (IU/L)
glucometabolic parameters | 6 months after the treatment
  alanine aminotransferase (IU/L)
glucometabolic parameters | 6 months after the treatment
  glycated hemoglobin (%)
glucometabolic parameters | 6 months after the treatment
  glycoalbumin (%)
glucometabolic parameters | 6 months after the treatment
  triglyceride (mg/dL)
glucometabolic parameters | 6 months after the treatment
  low-density lipoprotein (mg/dL)
glucometabolic parameters | 6 months after the treatment
  high-density lipoprotein (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of Internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided